CLINICAL TRIAL: NCT01249170
Title: Communication Skills Training and Competency Assessment for Pulmonary and Critical Care Medicine Fellows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer McCallister MD (Other)
Responsible Party: Sponsor-Investigator, Jennifer McCallister MD, Assistant Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010B0299
Record Dates: First submitted 2010-11-16; First posted 2010-11-29 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Communication
Keywords: Communication skills
MeSH Terms: conditions — Communication | interventions — Case-Control Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First year fellow (Other)
  Interventions: Behavioral: First year program
- Second Year Fellow (Other)
  Interventions: Other: Control comparison

INTERVENTIONS:
Behavioral: First year program — Information on group that underwent new educational program
  Arms: First year fellow
Other: Control comparison — Information from group that did not undergo new first year program
  Arms: Second Year Fellow

SUMMARY:
Study to determine if pulmonary/critical care fellows will demonstrate increased competency in the behavioral skills necessary to facilitate family meetings focused on discussions of goals of care in the ICU from pre- to post-communication skills training.

DETAILED DESCRIPTION:
The investigators hypothesize that pulmonary/critical care fellows will demonstrate increased competency in the behavioral skills necessary to facilitate family meetings focused on discussions of goals of care in the ICU from pre- to post-communication skills training.

ELIGIBILITY:
Inclusion Criteria:

* First- and second-year pulmonary/critical care fellows

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Subject self evaluation of training and skill | Measured at basline (Month 0)
  Determine level of prior training in communication skills and assess trainee attitudes about goals of care communication training

SECONDARY OUTCOMES:
Self versus trainer comparison assessment | Measured at basline (Month 0), during intervention and End of Study (Month 12)
  Compare pulmonary/critical care fellows' self-report of confidence and competence in performing goals of care discussions during family meetings with faculty observed competence in performance of this skill.
Evaluation of Effectiveness of intervention | Measured at End of Study (Month 12)
  Evaluate the effectiveness of a behavioral skills checklist as a formative feedback tool to improve the ability of pulmonary/critical care fellows to utilize the five key elements of patient-centered communication
Evaluate communication skills curriculum | Measured at End of Study (Month 12)
  Determine the effect of the implementation of a communication skills curriculum for pulmonary/critical care fellows on the physician communication domain of family satisfaction survey scores in the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McCallister, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States